CLINICAL TRIAL: NCT05979428
Title: A Phase I, Randomised, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0491-6075 Following Single Dose Administration to Healthy Participants and Multiple Doses to Participants With Dyslipidaemia
Brief Title: A Study to Look at How Safe a New Medicine (NNC0491-6075) is in Healthy People and in Participants With High Levels of Fat in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6491-4973; U1111-1285-1575 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers; Dyslipidaemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A Single ascending dose (SAD) cohorts in healthy participants: (Experimental): Healthy participants, randomized in 3:1 ratio in each of the cohorts will receive single ascending dose of either NNC0491-6075 or placebo in 5 cohorts (Cohort A1, A2, A3, A4 and A5). In cohorts A1, A2 and A3, the participants will receive subcutaneous injection, whereas in cohorts A4 and A5 the administration will be performed intravenously.
  Interventions: Drug: NNC0491-6075; Drug: Placebo
- Part B Multiple ascending dose (MAD) cohorts in dyslipidemia participants (Experimental): Participants with dyslipidemia, randomized in the ratio 2:1 in each of the cohorts will receive multiple ascending dose of either NNC0491-6075 or placebo in 3 cohorts (Cohort B1,B2 and B3). Participants will receive subcutaneous injections of either NNC0491-6075 or placebo once weekly for 4 weeks.
  Interventions: Drug: NNC0491-6075; Drug: Placebo
- Part C: Single ascending dose (SAD) cohorts in healthy Japanese participants: (Experimental): Healthy Japanese participants, randomized in the ratio 3:1 in each of the cohorts will receive single ascending dose of either NNC0491-6075 or placebo in 3 cohorts (Cohort C1,C2 and C3). The route of administration will be subcutaneous or intravenous.
  Interventions: Drug: NNC0491-6075; Drug: Placebo

INTERVENTIONS:
Drug: NNC0491-6075 — NNC0491-6075 will be administered as a subcutaneous injection in a skinfold in the abdomen or intravenously into a vein in the wrist, elbow, or the back of the hand.
Drug: Placebo — Placebo matched to NNC0491-6075 will be administered as a subcutaneous injection in a skinfold in the abdomen or intravenously into a vein in the wrist, elbow, or the back of the hand.

SUMMARY:
The study is testing a new study medicine to treat people with high levels of fat in the blood. The main aim of the study is to see if the new study medicine is safe and how it works in the body. Participants will either get NNC0491-6075 (the new study medicine) or placebo (a "dummy medicine" without active ingredients). Which treatment participants get is decided by chance. NNC0491-6075 is a new medicine which cannot be prescribed by doctors. The study has 3 parts (Part A, Part B and Part C). In Part A, investigators look at the effect of the study medicine after a single dose in healthy participants. Participants will get the study medicine either as injection(s) under the skin or as an infusion into a vein by the study staff. In Part B, investigators look at the effect of receiving the study medicine once weekly for four weeks in participants with high levels of fat in the blood but who are otherwise healthy. Participants will get the study medicine as injections under the skin by the study staff. In Part C, investigators look at the effect of the study medicine after a single dose in healthy participants of Japanese origin. Participants will get the study medicine either as injection(s) under the skin or as an infusion into a vein by the study staff. The study will last for about 18 months in total for Part A, Part B and Part C. Participants in Part A and Part C will be in the study for about 139 days each, from screening to the final visit while in Part B they will be in the study for about 160 days from screening to the final visit.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Men or women of non-childbearing potential
* Aged 18-55 years (both inclusive) at the time of signing informed consent
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests (presence of dyslipidaemia [example hypertriglyceridemia] is allowed) performed during the screening visit, as judged by the investigator
* Body mass index (BMI) between 18.5 and 34.9 kilograms per square meter (kg/m^2) (both inclusive) at screening
* Non-Japanese defined as not meeting inclusion criteria for Part C

Part B:

* Men or women of non-childbearing potential
* Aged 18-64 years (both inclusive) at the time of signing informed consent
* Dyslipidaemia at screening defined as all the below: Fasting serum triglycerides (TGs) greater than or equal to 150 milligrams per deciliter (mg/dL) and less than or equal to 500 mg/dL. Participants must have two measurements performed for eligibility. Both measurements must be greater than or equal to 135 mg/dL and at least one must be greater than or equal to 150 mg/dL. One of the measurements may be based on medical records or pre-screening results if the test is no more than 90 days old. If TGs are measured twice during the screening period, the tests must be performed with at least 4 days apart. TGs measured in the screening period must be after a 10 hour fast
* Fasting low-density lipoprotein cholesterol (LDL-C) greater than or equal to 50 mg/dL and less than 190 mg/dL
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator
* BMI between 18.5 and 34.9 kg/m^2 (both inclusive) at screening
* If on statin therapy the dose must have been stable for at least 8 weeks before screening and must be intended to remain stable throughout the study

Part C:

* Men or women of non-childbearing potential
* Aged 18-55 years (both inclusive) at the time of signing informed consent
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests (presence of dyslipidaemia [example, hypertriglyceridemia] is allowed) performed during the screening visit, as judged by the investigator
* BMI between 18.5 and 34.9 kg/m^2 (both inclusive) at screening
* Japanese defined as both biological parents of Japanese descent

Exclusion Criteria:

Part A,B and C:

* Known or suspected hypersensitivity to study intervention(s) or related products
* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* Use of prescription or non-prescription medicinal products within 14 days before screening. Exceptions are: Topical medications; occasional use of over-the-counter acetaminophen or Non-steroidal anti-inflammatory drugs (NSAIDs) at their labelled doses for mild pain; and statin therapy in Part B only if the dose has been stable for at least 8 weeks prior to screening and is intended to remain stable throughout the trial
* Any laboratory safety parameters at screening outside the below laboratory ranges, see designated reference range documents for specific values: Alanine aminotransferase greater than upper limit of normal (ULN) +50 percentage (%), Aspartate aminotransferase greater than ULN +50%, Total Bilirubin greater than ULN +20%, Creatine kinase greater than ULN +50%.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Part A (SAD): Number of treatment emergent adverse events (TEAEs) | From pre-dose (Day 1) to end of study (Day 110)
  Measured as count of events. An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. A TEAE is defined as an AE that either has onset time after first trial product administration and no later than the end of study visit or Is present before first trial product administration and increases in severity during the treatment period and no later than the end of study visit.
Part B (MAD): Number of treatment emergent adverse events (TEAEs) | From pre-dose (Day 1) to end of study (Day 131)
  Measured as count of events. An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. A TEAE is defined as an AE that either has onset time after first trial product administration and no later than the end of study visit or Is present before first trial product administration and increases in severity during the treatment period and no later than the end of study visit.
Part C (SAD): Number of treatment emergent adverse events (TEAEs) | From pre-dose (Day 1) to end of study (Day 110)
  Measured as count of events. An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. A TEAE is defined as an AE that either has onset time after first trial product administration and no later than the end of study visit or Is present before first trial product administration and increases in severity during the treatment period and no later than the end of study visit.

SECONDARY OUTCOMES:
Part A (SAD): AUC0-∞, SD; the area under the NNC0491-6075 serum concentration-time curve from 0 to infinity after a single dose | From pre-dose (Day 1) to end of study (Day 110)
  Measured as hours*nanomoles per liter (h*nmol/L)
Part A (SAD): Cmax, SD; the maximum serum concentration of NNC0491-6075 after a single dose | From pre-dose (Day 1) to end of study (Day 110)
  Measured as nanomoles per liter (nmol/L)
Part A (SAD): t½, SD; the terminal half-life of NNC0491-6075 after a single dose | From pre-dose (Day 1) to end of study (Day 110)
  Measured as hours (h)
Part A (SAD): tmax, SD; The time to maximum concentration of NNC0491-6075 after a single-dose (only from subcutaneous administration) | From pre-dose (Day 1) to end of study (Day 110)
  Measured as hours
Part B (MAD): AUC0-168h, MD; the area under the NNC0491-6075 serum concentration-time curve from time 0 to 168 hours after last dose | From pre-dose (Day 22) to 168 hours after last dose (Day 29)
  Measured as h*nmol/L
Part B (MAD): Cmax, MD; the maximum serum concentration of NNC0491-6075 after last dose | From pre-dose (Day 22) to end of study (Day 131)
  Measured as nmol/L
Part B (MAD): t½, MD; the terminal half-life of NNC0491-6075 after last dose | From pre-dose (Day 22) to end of study (Day 131)
  Measured as hours
Part B (MAD): tmax, MD; The time to maximum concentration of NNC0491-6075 after last dose | From pre-dose (Day 22) to end of study (Day 131)
  Measured as hours
Part C (SAD): AUC0-∞, SD; the area under the NNC0491-6075 serum concentration-time curve from 0 to infinity after a single dose | From pre-dose (Day 1) to end of study (Day 110)
  Measured as h*nmol/L
Part C (SAD): Cmax, SD; the maximum serum concentration of NNC0491-6075 after a single dose | From pre-dose (Day 1) to end of study (Day 110)
  Measured as nmol/L
Part C (SAD): t½, SD; the terminal half-life of NNC0491-6075 after a single dose | From pre-dose (Day 1) to end of study (Day 110)
  Measured as hours
Part C (SAD): tmax, SD; The time to maximum concentration of NNC0491-6075 after a single-dose (only from subcutaneous administration) | From pre-dose (Day 1) to end of study (Day 110)
  Measured as hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical LA, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com